CLINICAL TRIAL: NCT03880188
Title: Fat to the Future, Dermal Time 2: Long Term Clinical and Histological Status of Free Dermal Fat Autograft Recipient Sites: Cross-Sectional Assessment in a Retrospective Cohort Treated for Complex Craniofacial Wounds
Brief Title: Long Term Status of Free Dermal Fat Autografts for Complex Craniofacial Wounds
Acronym: FTFDT2
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dufresne, Craig, MD, PC (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1219-3733; 000083 (Other: FSRG #1 IRB)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Wounds and Injuries; Wound Infection; Facial Bones Fracture; Soft Tissue Injuries; Skull Fractures; Surgical Wound; Surgical Wound Infection; Wound Healing; Disturbance of Wound Healing; Wound; Head, Multiple; Wound; Head, Scalp; Wound; Head; Wound Complication; Wound Dehiscence; Wound of Skin; Wound Open; Wounds, Penetrating; Wounds, Nonpenetrating; Wounds
Keywords: Autologous Transplantation; Free Tissue Flaps; Graft Survival; Reconstructive Surgical Procedures; Patient Selection; Debridement; Subcutaneous Fat; Surgical Flaps; Treatment Outcome
MeSH Terms: conditions — Wounds and Injuries; Wound Infection; Soft Tissue Injuries; Skull Fractures; Surgical Wound; Surgical Wound Infection; Wounds, Penetrating; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Prepared and stained slides made from the material obtained during biopsies will be retained for use in the clinical care of the patient and research. Other material stored in formalin from biopsy specimens obtained will be banked for future use in immunohistochemistry studies to further define free DFA physiology. Additional IRB approval to use any the material from biopsy specimens for any future studies will be obtained. The specimens will not be shared with outside researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the use of free autologous dermal fat grafting (also called free dermal fat autografting) to treat complex craniofacial wounds that have failed standard treatment and to understand how well these grafts work to repair wounds long term. Patients who have undergone free autologous dermal fat grafting to treat complex craniofacial wounds 2-30 years ago will have photographs and small biopsies taken of the area that was grafted.

DETAILED DESCRIPTION:
Complex craniofacial wounds (CCW) are those considered to be refractory to initial reconstructive and antibiotic treatment and may involve chronic infection, exposed hardware, irradiated local tissue, and soft tissue volume loss. They are a functional, aesthetic, quality-of-life, and economic burden and have many aetiologies and impact patients of all ages from diverse socio-economic and geographical backgrounds. The present study will evaluate if free dermal fat autografts (DFA) can serve as a less involved, more dynamic approach than the standard of microvascular flaps to facilitate healing and reconstruction for CCW. A previous 33-year retrospective study of free DFA for CCW indicated recipient graft sites healed and remained volume-stable in most patients. To evaluate the long-term viability of this modality, clinical and histological assessments of free DFA recipient and undisturbed tissue at donor sites will be carried out in patients from the original cohort. In the present study, it will be first determined if free DFA continues to provide stable long-term outcomes for prevention of infection and hardware exposure and stable volume and contour results. Then, it will be determined if free DFA recipient sites retain normal, expected histology and immune cells (dermal lymphocytes, macrophages, and mast cells). Finally, it will be evaluated if the long-term free DFA recipient site tissues are significantly different from undisturbed tissue at donor sites with respect to the presence of adipose tissue and populations of immune cells. The present study will be the first to (1) evaluate the long-term fate of free DFA recipient sites in this complex craniofacial wounds, (2) determine the presence of immune cells within free DFA recipient sites, and (3) compare the long-term differences of free DFA recipient and undisturbed tissue at donor sites. Outcomes from this project will serve as the basis of understanding of free DFA survival and function in treating CCW and provide an investigative framework for more rigorous follow-up studies to define indications and refine techniques for free DFA use in this context and more generally.

ELIGIBILITY:
Inclusion Criteria:

* Underwent free autologous dermal fat grafting carried out by the Study Principal Investigator for one or more complex craniofacial wounds
* Speaks, reads, and understands English
* Willing to freely give consent
* Is able or has a legal representative to give consent

Exclusion Criteria:

* Did not have free autologous dermal fat grafting
* Did not undergo free autologous dermal fat grafting carried out by the Study Principal Investigator
* Underwent free autologous dermal fat grafting carried out by the Study Principal Investigator for an indication other than for one or more complex craniofacial wounds
* Lacks sufficient chart data for study requirements
* Patients for whom it cannot be determined when they underwent free vs injected autologous dermal fat grafting
* Does not speak, read, or understand English
* Unwilling to freely give consent
* Is unable or does not have a legal representative to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential patients are drawn from a retrospective cohort of consecutive patients who underwent free autologous dermal fat grafting for one or more complex craniofacial wounds between 1985 and 2018, carried out by a single sub-speciality trained plastic surgeon (Study Principal Investigator).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing and defect amelioration. | Outcomes are evaluated at one clinical encounter, lasting approximately 1 hour.
  Wound healing and defect amelioration will be clinically evaluated. Evaluation will be based on the absence of drainage, erythema, and oedema; reduction of pain; the presence of intact tissues and stable volume and contour in the area where the graft was placed.

SECONDARY OUTCOMES:
Histology and the presence of stem and immune cells in the free autologous dermal fat graft recipient site. | Outcomes are evaluated at one clinical encounter, lasting approximately 1 hour.
  Histology and the presence of stem and immune cells in the free autologous dermal fat graft recipient site will be qualitatively and quantitatively evaluated, according to standard laboratory procedures of the receiving institution, using the biopsies taken during the consultation and minor procedure visit.
Histology and the presence of stem and immune cells in the native local tissue. | Outcomes are evaluated at one clinical encounter, lasting approximately 1 hour.
  Histology and the presence of stem and immune cells in the native local tissue will be qualitatively and quantitatively evaluated, according to standard laboratory procedures of the receiving institution, using the biopsies taken during the consultation and minor procedure visit.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Dufresne, MD, Principal Investigator — Dr Craig R Dufresne, MD, PC
Locations (1):
- Office of Craig R Dufresne, MD, PC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) or biospecimens will be shared.

REFERENCES:
- [Background] Dufresne CR, Poling MI. Free Dermal Fat Autografting for Complex Craniofacial Wounds. J Craniofac Surg. 2020 Sep;31(6):1563-1567. doi: 10.1097/SCS.0000000000006398. PMID 32310868
- [Background] Dufresne CR, Poling MI. Free Dermal Fat Autografts for Complex Craniofacial Wounds: A 3-decade, Retrospective Cohort Study. PRS Global Open. 2019 August; 7(8S-1):101. doi: 10.1097/01.GOX.0000584800.01063.18.
- See also: Principal Investigator's (Dr Craig R Dufresne) Research and Press Relations main webpage. Last Accessed: 7 Jun 2022 — https://www.duplastics.com/research-press/